CLINICAL TRIAL: NCT01831154
Title: The Effect of Intraoperative Tight Glycemic Control on Surgical Site Infection Rates in Patients Undergoing Open Heart Surgery
Brief Title: The Effect of Tight Glycemic Control on Surgical Site Infection Rates in Patients Undergoing Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Collaborators: University of South Florida (Other)
Responsible Party: Principal Investigator, Sierra Gower, Dr., James A. Haley Veterans Administration Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 106219
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Hyperglycemia; Surgical Site Infection
Keywords: Glycemic control
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tight Glycemic Group (Experimental): The tight glycemic group received a continuous intravenous infusion of regular insulin in the intraoperative period titrated per a modified Portland Protocol from Vanderbilt University Medical Center, Tennessee. The initial bolus of insulin and insulin infusion was initiated prior to induction of anesthesia if the morning blood glucose was greater than 149 mg/dl or any time intraoperatively the blood glucose elevated above 149 mg/dl.The titration of insulin for the tight glycemic group maintained blood glucose levels between 110-149 mg/dl throughout the intraoperative period. The intraoperative blood glucose was titrated to blood glucose levels sampled every 30 minutes.Upon transfer to the intensive care unit the protocol ended and all subjects received the same glycemic control.
  Interventions: Drug: Tight Glycemic
- Conventional Glycemic Group (Experimental): The conventional glycemic group received a continuous intravenous infusion of regular insulin in the intraoperative period titrated per a modified Portland Protocol from Vanderbilt University Medical Center, Tennessee. The initial insulin bolus and infusion was initiated prior to induction of anesthesia if the morning blood glucose was greater than 180 mg/dl or any time intraoperatively that the blood glucose elevated above 180 mg/dl. The insulin infusion was titrated throughout the intraoperative period to maintain blood glucose levels between 150-180 mg/dl.The intraoperative blood glucose was titrated to blood glucose levels sampled every 30 minutes. Upon transfer to the ICU the intraoperative protocol ended and all subjects received the standardized glycemic control for the ICU.
  Interventions: Drug: Conventional Glycemic
- Standard Glycemic Group (Experimental): The standard glycemic group received intravenous injections of regular insulin in the intraoperative period titrated per the usual care protocol utilized at the study site. The initial bolus of insulin was initiated prior to induction of anesthesia if the morning blood glucose is greater than 180 mg/dl or any time intraoperatively that the blood glucose rises above 180 mg/dl. The intraoperative blood glucose was titrated to blood glucose levels sampled every 30 minutes.Upon transfer to the ICU the intraoperative protocol ended and all subjects received the standardized glycemic control for the ICU.
  Interventions: Drug: Standard Glycemic

INTERVENTIONS:
Drug: Tight Glycemic — The insulin infusion consisted of 100 units of regular insulin in 100 ml of normal saline.
  Arms: Tight Glycemic Group
Drug: Conventional Glycemic — The insulin infusion consisted of 100 units of regular insulin in 100 ml of normal saline.
  Arms: Conventional Glycemic Group
Drug: Standard Glycemic — Insulin was Regular Insulin administered intravenous bolus.
  Arms: Standard Glycemic Group

SUMMARY:
The purpose of this study was to investigate the effects of three different glycemic treatment conditions (tight, conventional, and standard) in the intraoperative period on: 1) postoperative surgical site infections, and 2) postoperative procalcitonin, and C-reactive protein levels in patients undergoing open-heart surgery. Secondary aims of the study were to investigate the effects of the three glycemic treatment conditions on: 1) intraoperative blood glucose; 2) intraoperative glycemic stability; and 3) intensive care unit length of stay, in patients undergoing open-heart surgery.

DETAILED DESCRIPTION:
An experimental design with a multilevel, single factor, within-subjects design was utilized. Patients were nested within anesthesia provider teams. The design was counterbalanced by means of a Latin square, where each of three anesthesia provider teams dispensed each of three glycemic treatment conditions once.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 21
* on cardiopulmonary bypass or off cardiopulmonary
* elective or urgent coronary artery bypass graft (CABG) surgery
* CABG with or without combined valve surgery
* valve surgery

Exclusion Criteria:

* chronically immunosuppressed
* suffered from end-stage organ disease
* currently had active infections
* underwent emergent or salvage CABG surgery
* had an implanted insulin pump
* were in another interventional clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sierra A Gower, PhD, Principal Investigator — James A Haley VAH; Theresa Beckie, PhD, Study Chair — University of South Florida
Locations (1):
- James A. Haley VAH, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Started | 15 (Study Institutional Review Board (IRB) approval 11-11-2009, first subjects enrolled 6-7-2010) | 11 (Study IRB approval 11-11-2009, first subjects enrolled 6-7-2010) | 11 (Study IRB approval 11-11-2009, first subjects enrolled 6-7-2010)
Completed | 15 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group | Total
Number analyzed (Participants) | 15 | 11 | 11 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.9) | 66 (7.4) | 66 (4) | 65 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 15 | 11 | 11 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 14 | 9 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 15 | 11 | 10 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 11 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Undergoing Open Heart Surgery With Postoperative Surgical Site Infection
Description: The presence or absence of deep, or/and superficial sternal wound infection and deep, superficial harvest site infection within in six weeks postoperatively was a primary outcome variable. Infection assessment was performed during the intensive care phase, at hospital discharge, two-week post hospital discharge and six-week post hospital discharge by independent blinded researchers that were part of the cardiothoracic team.
Time Frame: six weeks postoperatively
Population: Inclusion > age 21, underwent elective or urgent Coronary Artery Bypass Graft (CABG) with or without combined valve surgery or valve surgery alone, on or off cardiopulmonary bypass (CPB). Exclusions were patients diagnosed with immunosuppression, end stage organ disease, or active infections.
Measure: Number; unit: participants
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Number analyzed (Participants) | 15 | 11 | 11
participants | 4 | 5 | 5
Statistical Analysis 1: Comparison: Tight Glycemic Group vs Conventional Glycemic Group vs Standard Glycemic Group; Cross tabulation with statistical testing with chi-square and Cramer's V was performed on infection to determine if there was any difference in surgical site infections between the interventional groups in 30 day period; Test type: Superiority or Other; p = 0.512, Chi-squared; Chi-squared value of 1.34 and Cramer's V .190

2. Primary Outcome: The Effect of Intraoperative Tight Glycemic Control on Postoperative Procalcitonin Plasma Levels in Patients Undergoing Open Heart Surgery
Description: Procalcitonin concentrations were collected in addition to clinical signs for indications of infection. These biomarker concentrations were collected after successful separation from cardiopulmonary bypass (CPB), and every morning for five days postoperatively. Values were drawn by anesthesia providers and intensive care unit (ICU) registered nurses or laboratory personnel with the standard morning blood work. All procalcitonin blood values from post cardiopulmonary bypass through postoperative day 5 were collected. The outcome measure was mean procalcitonin values with standard deviation.
Time Frame: Post CPB and Postoperative days 1 through 5
Population: Inclusion > age 21, underwent elective or urgent CABG with or without combined valve surgery or valve surgery alone, on or off CPB. Exclusions were patients diagnosed with immunosuppression, end stage organ disease, or active infections. Six participants had > 50% missing data and were dropped from this analysis (4 tight, 1 in other two groups).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Number analyzed (Participants) | 11 | 10 | 10
ng/ml | 0.466 (0.448) | 1.15 (0.981) | 1.082 (0.581)
Statistical Analysis 1: Comparison: Tight Glycemic Group vs Conventional Glycemic Group vs Standard Glycemic Group; Test type: Superiority or Other; p = 0.024, ANOVA

3. Primary Outcome: The Effect of Intraoperative Tight Glycemic Control on Postoperative C-Reactive Protein Plasma Levels in Patients Undergoing Open Heart Surgery
Description: C-Reactive Protein concentrations were collected in addition to clinical signs for indications of infection. These biomarker concentrations were collected after successful separation from cardiopulmonary bypass (CPB), and every morning for five days postoperatively. Values were drawn by anesthesia providers and intensive care unit (ICU) registered nurses or laboratory personnel with the standard morning blood work. All C-Reactive Protein blood values from post cardiopulmonary bypass through postoperative day 5 were collected. The outcome measure was mean C-Reactive Protein values with standard deviation.
Time Frame: Post cardiopulmonary bypass and postoperative day 1 through 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Mg/L
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Number analyzed (Participants) | 11 | 10 | 10
Mg/L | 13.11 (3.52) | 10.95 (3.48) | 13.98 (4.22)

4. Secondary Outcome: Intraoperative Blood Glucose Levels in Patients Undergoing Open Heart Surgery
Description: Blood glucose values were obtained every 30 minutes in the intraoperative period, and were drawn and recorded by the certified registered nurse anesthetist (CRNA) performing the anesthetic. Repeated measured ANOVA with Greenhouse-Geisser correction was employed to determine if participants assigned to the tight glycemic group yielded lower blood glucose levels intraoperatively (every 30 minutes for 240 minutes) than the other two interventions. All blood glucose measures over the intraoperative period were averaged to produce a mean and standard deviation comparing the tight glycemic group to the other two interventional groups, Data points were blood glucose testing collected every 30 minutes starting on entry into the operating room.
Time Frame: Blood glucose measured every 30 minutes starting on entry into the operating room until exiting the operating room or 240 minutes, whichever event occurred first
Population: Inclusion > age 21, underwent elective or urgent CABG with or without combined valve surgery or valve surgery alone, on or off CPB. Exclusions were patients diagnosed with immunosuppression, end stage organ disease, or active infections.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Number analyzed (Participants) | 15 | 11 | 11
mg/dl | 130.77 (22.04) | 143.33 (29.59) | 145.55 (35.15)
Statistical Analysis 1: Comparison: Tight Glycemic Group vs Conventional Glycemic Group vs Standard Glycemic Group; Test type: Superiority or Other; p = 0.132, ANOVA

5. Secondary Outcome: The Effect of Tight Glycemic Control on Intensive Care Unit Length of Stay in Patients Undergoing Open Heart Surgery
Description: Length of stay (LOS) in the intensive care unit was measured by the total number of days each patient stayed in the intensive care unit.
Time Frame: ICU days measured every day the patient stayed in ICU starting with entry into the ICU from the Operating Room until discharge from the ICU to the ward
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Number analyzed (Participants) | 15 | 11 | 11
days | 7 (5.29) | 6.18 (4.9) | 7.18 (6.03)
Statistical Analysis 1: Comparison: Tight Glycemic Group vs Conventional Glycemic Group vs Standard Glycemic Group; Test type: Superiority or Other; p = 0.908, ANOVA — A one way ANOVA was used to determine if participants in the tight glycemic group had shorter intensive care unit (ICU) length of stay (LOS) than participants in the other interventional groups

6. Secondary Outcome: Intraoperative Glycemic Stability in Patients Undergoing Open Heart Surgery Compared Between Three Glycemic Protocols.
Description: Intraoperative glycemic stability was operationalize as how often blood glucose levels were maintained as normal or maintained in the preset target ranges for each group. If intraoperative blood glucose levels fell outside of normal (hypoglycemia or hyperglycemia) or, outside the preset target ranges, for each protocol, for 3 consecutive blood glucoses (1.5 hours) despite insulin therapy a marker of inadequate glycemic control was recorded.
Time Frame: Measures of blood glucose every 30 minutes starting on entry into the operating room until exiting the operating room or 240 minutes whichever event occurred first
Population: Inclusion > age 21, underwent elective or urgent CABG with or without combined valve surgery or valve surgery alone, on or off CPB. Exclusions were patients diagnosed with immunosuppression, end stage organ disease, or active infections. No data analysis could be performed because there were too few episodes of glycemic instability.
Measure: Number; unit: episodes out of target glucose range
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Number analyzed (Participants) | 15 | 11 | 11
episodes out of target glucose range | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: The study period including follow up was for 16 months in time, June 2010 through October 2011.
Arm/Group | Tight Glycemic Group | Conventional Glycemic Group | Standard Glycemic Group
Serious Adverse Events (participants affected / at risk) | 4/15 | 1/11 | 5/11
Other Adverse Events (participants affected / at risk) | 0/15 | 0/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tight Glycemic Group (N=15) | Conventional Glycemic Group (N=11) | Standard Glycemic Group (N=11)
Atrial Fibrillation (Cardiac disorders) | 2 (4) | 1 (4) | 1 (4)
Cerebral vascular accident (CVA) (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2)
Deep sternal wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Chest pain, restenosis of cardiac bypass graft
Feet Ulcerations (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Bilateral Feet blisters and ulceration
Viral gastrointestinal-dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Peripheral edema, dyspnea, fluid overload
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) — death

LIMITATIONS AND CAVEATS:
This study was conducted in a single center and homogenous sample. Statistical power was not sufficient to draw conclusion on the effect of tight glycemic control on postoperative outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No